CLINICAL TRIAL: NCT02791282
Title: CHANGE-MRI (CTEPH DIAGNOSIS Europe - MRI)
Brief Title: CTEPH DIAGNOSIS Europe - MRI
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hannover Medical School (Other)
Collaborators: University of Sheffield (Other); University of Giessen (Other); Ludwig-Maximilians - University of Munich (Other); Heidelberg University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHANGE-MRI
Record Dates: First submitted 2016-06-01; First posted 2016-06-06 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-06

CONDITIONS: Pulmonary Hypertension
Keywords: Chronic Thromboembolic Pulmonary Hypertension (CTEPH); MRI; SPECT
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Index test: functional dynamic contrast enhanced (DCE)-MRI (Other): Patients with clinical suspicion for CTEPH, scheduled for SPECT
  Interventions: Other: Index test: functional dynamic contrast enhanced (DCE)-MRI

INTERVENTIONS:
Other: Index test: functional dynamic contrast enhanced (DCE)-MRI — Index test: functional dynamic contrast enhanced (DCE)-MRI Reference test: Ventilation-perfusion (VQ) single-photon emission computed tomography (SPECT) Follow-up per patient: clinical assessment after 6-12 months

SUMMARY:
Phase III diagnostic trial to demonstrate that functional lung MRI can replace VQ-SPECT in a diagnostic strategy for patients with suspected CTEPH where positive findings are verified with catheter pulmonary angiography (CPA), or computed tomography pulmonary angiography (CTPA)

DETAILED DESCRIPTION:
CHANGE-MRI is a prospective, multicentre, comparative phase III diagnostic study. The study aims to show via an in-place validation that MRI can replace VQ-SPECT as a screening test for chronic pulmonary embolism in the diagnostic algorithm for CTEPH. The diagnostic gold standard is catheter pulmonary angiography (CPA) or computed tomography pulmonary angiography (CTPA) with correction from the clinical outcome after 6-12 months.

ELIGIBILITY:
Inclusion Criteria:

* Transthoracic echocardiography indicates pulmonary hypertension
* Patients with clinical suspicion for CTEPH, scheduled for SPECT
* Provided informed consent for the study
* Age >18y

Exclusion Criteria:

* Patient unable to undergo MRI (e.g. due to claustrophobia, cardiac pacemaker, hypersensitivity to MR i.v. contrast imaging agents)
* Women who are pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1080 (Estimated)
Dates: Start 2016-05; Primary Completion 2020-03 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with positive MRI in the group of patients who have a positive VQ-SPECT diagnosis for chronic pulmonary embolism and who are positive in the gold standard | 6 months
The proportion of patients with positive MRI in the group of patients with negative VQ-SPECT who are negative in the gold standard | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jens Vogel-Claussen, MD, Principal Investigator — Hannover Medical School
Locations (1):
- Hannover Medical School, Hanover, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lasch F, Karch A, Koch A, Derlin T, Voskrebenzev A, Alsady TM, Hoeper MM, Gall H, Roller F, Harth S, Steiner D, Krombach G, Ghofrani HA, Rengier F, Heussel CP, Grunig E, Beitzke D, Hacker M, Lang IM, Behr J, Bartenstein P, Dinkel J, Schmidt KH, Kreitner KF, Frauenfelder T, Ulrich S, Hamer OW, Pfeifer M, Johns CS, Kiely DG, Swift AJ, Wild J, Vogel-Claussen J. Comparison of MRI and VQ-SPECT as a Screening Test for Patients With Suspected CTEPH: CHANGE-MRI Study Design and Rationale. Front Cardiovasc Med. 2020 Apr 9;7:51. doi: 10.3389/fcvm.2020.00051. eCollection 2020. PMID 32328500
- See also: study website — http://change-mri.de